CLINICAL TRIAL: NCT06899659
Title: A Prospective Multi-Center, Randomized Controlled Pre-Market Clinical Trial to Assess the Safety and Effectiveness of the JuggerStitch™ Meniscal Repair Device for Arthroscopic Meniscal Repair
Brief Title: Evaluation on Safety and Effectiveness of the An All-inside, All-suture Meniscal Repair Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Huashan Hospital (Other); Hunan Provincial People's Hospital (Other); Wuhan TongJi Hospital (Other); First Affiliated Hospital of Jinan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEA2020-26SM
Record Dates: First submitted 2025-02-19; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Meniscal Tears
Keywords: Meniscal Repair; Arthroscopic Surgery; JuggerStitch™ Meniscal Repair Device

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: the investigational group (JuggerStitch™ Meniscal Repair Device) or the control group (Fast-Fix 360 Meniscal Repair System).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Investigational Group (Experimental): Participants in this group will receive the JuggerStitch™ Meniscal Repair Device for arthroscopic meniscal repair. The JuggerStitch™ device is a new all-inside meniscal repair system that consists of a suture device and various auxiliary tools. It is designed to repair vertical longitudinal full-thickness tears (e.g., bucket-handle) in the red-red and red-white zones of the meniscus.
  Interventions: Device: JuggerStitch™ Meniscal Repair Device
- Control Group (Experimental): Participants in this group will receive the Fast-Fix 360 Meniscal Repair System for arthroscopic meniscal repair. The Fast-Fix 360 is a well-established all-inside meniscal repair device that consists of a suture and two fixed rods. It is designed to repair meniscal tears in a similar manner to the JuggerStitch™ device.
  Interventions: Device: Fast-Fix 360 Meniscal Repair System

INTERVENTIONS:
Device: JuggerStitch™ Meniscal Repair Device — Participants assigned to investigational group undergoing arthroscopy meniscal repair with JuggerStitch™ Meniscal Repair Device.
  Arms: Investigational Group
Device: Fast-Fix 360 Meniscal Repair System — Participants assigned to control group undergoing arthroscopy meniscal repair with the Fast-Fix 360 Meniscal Repair System.
  Arms: Control Group

SUMMARY:
This study is a prospective, multi-center, randomized controlled pre-market clinical trial in China to evaluate the safety and efficacy of the JuggerStitch™ Meniscal Repair Device for arthroscopic meniscal repair. The study aims to compare the clinical outcomes of the JuggerStitch™ device with the Fast-Fix 360 Meniscal Repair System in patients with meniscal tears. The primary endpoint is the Lysholm Knee Score at 6 months postoperatively, and secondary endpoints include immediate device success rate, Tegner Activity Score, Visual Analogue Scale (VAS) score for pain, meniscal healing evaluated by MRI, and device-related adverse event rate. The study will enroll 94 subjects across 5 clinical sites.

DETAILED DESCRIPTION:
1. Purpose of the Study The purpose of this study is to evaluate the safety and efficacy of the JuggerStitch™ Meniscal Repair Device for arthroscopic meniscal repair in patients with meniscal tears. The study will compare the clinical outcomes of the JuggerStitch™ device with the Fast-Fix 360 Meniscal Repair System, a well-established device for meniscal repair.
2. Study Design and Methodology This is a prospective, multi-center, randomized controlled pre-market clinical trial. The study will involve 5 clinical sites and will enroll a total of 94 subjects. Subjects will be randomly assigned to either the investigational group (JuggerStitch™ device) or the control group (Fast-Fix 360 device). The primary endpoint is the Lysholm Knee Score at 6 months postoperatively, and secondary endpoints include immediate device success rate, Tegner Activity Score, VAS score for pain, meniscal healing evaluated by MRI, and device-related adverse event rate.
3. Inclusion and Exclusion Criteria 1) Inclusion Criteria: Age between 18 and 60 years; Scheduled for meniscal repair with a vertical longitudinal full-thickness tear (e.g., bucket-handle) in the red-red and red-white zones; Able to understand all risks and benefits described in the informed consent form and willing to comply with the rehabilitation and follow-up visits specified in the clinical trial protocol.

2) Exclusion Criteria: Meniscal tears in the avascular zone of the meniscus; Meniscal tears not suitable for repair due to the degree of damage (marked irregularity and complex tearing) to the meniscus body, including degenerative, radial, horizontal cleavage, flap, and root tears; Multiple ligament injuries of the affected knee joint; Adhesion of the affected knee joint; Planned intraoperative or postoperative intra-articular injection; Articular surface cartilage injury of the targeted knee assessed by the International Cartilage Repair Society (ICRS) is grade 3-4; Kellgren-Lawrence grades of documented radiographic evidence of osteoarthritis (OA) in the affected knee is ≥III; Instability or valgus/varus deformity (>5°) of the affected knee; Acute or chronic, local or systemic infections; Metabolic diseases; Abnormal liver and kidney function (creatinine 3 times higher than the upper limit of normal value or alanine aminotransferase or aspartate aminotransferase 3 times higher than the upper limit of normal value) before operation; History of operation in the affected knee; Acute myocardial infarction or stroke occurred within 6 months before operation; Known allergy to any material (polyethylene, polypropylene, polyester, polyetheretherketone) of the implants; Pregnant or known to be pregnant; Other circumstances that the researchers believe may affect the efficacy and safety evaluation of the investigated medical devices; Currently participating in other clinical trials;

4. Surgical Procedure The surgical procedure will involve arthroscopic exploration and repair of the meniscal tear using either the JuggerStitch™ device or the Fast-Fix 360 device. The specific steps for each device will be followed according to the manufacturer's instructions and the surgeon's standard operating procedures.

Postoperative Rehabilitation and Follow-up: Postoperative rehabilitation will include the use of an elastic bandage, appropriate massage to prevent blood clots, and guidance on quadriceps isometric contraction and straight leg-raising training. Subjects will be followed up at 3 months, 6 months, and 12 months postoperatively. At each follow-up visit, the Lysholm Knee Score, Tegner Activity Score, and VAS score for pain will be recorded. MRI of the knee joint will be performed at 6 months and 12 months postoperatively to evaluate meniscal healing.

Assessment of Efficacy and Safety: Efficacy will be assessed using the Lysholm Knee Score, Tegner Activity Score, and VAS score for pain. Safety will be assessed by monitoring and recording adverse events, including device-related adverse events, during the follow-up period.

Statistical Considerations: The sample size calculation is based on the difference in Lysholm Knee Score at 6 months postoperatively. A total of 94 subjects will be enrolled, with 47 subjects in each group. The primary endpoint will be analyzed using a covariance analysis model, and the secondary endpoints will be analyzed using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Scheduled for meniscal repair with a vertical longitudinal full-thickness tear (e.g., bucket-handle) in the red-red and red-white zones
* Able to understand all risks and benefits described in the informed consent form and willing to comply with the rehabilitation and follow-up visits specified in the clinical trial protocol

Exclusion Criteria:

* Meniscal tears in the avascular zone of the meniscus
* Meniscal tears not suitable for repair due to the degree of damage (marked irregularity and complex tearing) to the meniscus body, including degenerative, radial, horizontal cleavage, flap, and root tears
* Multiple ligament injuries of the affected knee joint
* Adhesion of the affected knee joint
* Planned intraoperative or postoperative intra-articular injection
* Articular surface cartilage injury of the targeted knee assessed by the - International Cartilage Repair Society (ICRS) is grade 3-4 Kellgren-Lawrence grades of documented radiographic evidence of osteoarthritis (OA) in the affected knee is ≥III
* Instability or valgus/varus deformity (>5°) of the affected knee
* Acute or chronic, local or systemic infections
* Metabolic diseases
* Abnormal liver and kidney function (creatinine 3 times higher than the upper limit of normal value or alanine aminotransferase or aspartate aminotransferase 3 times higher than the upper limit of normal value) before operation
* History of operation in the affected knee
* Acute myocardial infarction or stroke occurred within 6 months before operation
* Known allergy to any material (polyethylene, polypropylene, polyester, polyetheretherketone) of the implants
* Pregnant or known to be pregnant
* Other circumstances that the researchers believe may affect the efficacy and safety evaluation of the investigated medical devices
* Currently participating in other clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Lysholm Knee Score | Post-op 6 months
  The Lysholm Knee Score is a widely used and validated tool for assessing knee function, particularly in patients with meniscal injuries. It evaluates eight aspects of knee function: limp, use of cane or crutches, locking sensation, giving way sensation, pain, swelling, climbing stairs, and squatting. Each aspect is scored on a scale, and the total score ranges from 0 to 100, with higher scores indicating better knee function.

SECONDARY OUTCOMES:
Immediate Device Success Rate | Intraoperatively
  The immediate device success rate is defined as the proportion of successful sutures of the injured site without any additional instruments (except matching surgical tools) during the operation. It is calculated as the number of successfully implanted anchors divided by the total number of implanted anchors, multiplied by 100%.
Tegner Activity Score | Post-op 3, 6, and 12 months
  The Tegner Activity Score is a validated tool for assessing the level of physical activity in patients with knee injuries. It ranges from 0 (sick leave or disability pension because of knee problems) to 10 (competitive sports at a national elite level). The score is based on the highest level of activity the patient can participate in before and after the injury.
Visual Analogue Scale (VAS) Score for Pain | Post-op 3, 6, and 12 months
  The VAS is a validated tool for assessing pain intensity. It is a 10 cm horizontal line, where 0 represents no pain and 10 represents the worst possible pain. Patients mark the point on the line that corresponds to their pain level.
Meniscal Healing Evaluated by Magnetic Resonance Imaging (MRI) | Post-op 6 and 12 months
  MRI will be used to evaluate the healing of the meniscus at 6 and 12 months postoperatively. The MRI results will be classified according to the MRI classification for meniscal tear after arthroscopy repair, which ranges from Grade 0 (normal) to Grade III (high signal in the meniscus reaches the articular surface of the meniscus).

CONTACTS AND LOCATIONS:
Overall Officials: Shiyi Chen, MD, Principal Investigator — Huashan Hospital
Locations (2):
- China (2):
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No
The study does not currently have a plan to share individual participant data due to privacy and confidentiality concerns. The data may contain sensitive information that could potentially identify participants, and sharing it could compromise their privacy. Additionally, the study is subject to regulatory and ethical requirements that limit the sharing of individual participant data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT06899659/Prot_SAP_000.pdf